CLINICAL TRIAL: NCT04019769
Title: Phase 1 Trial of Glutamine Supplementation in Patients With Immune Dysregulation
Brief Title: Glutamine Supplementation in People With Immune Dysregulation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left NIH. No subjects enrolled.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190121; 19-I-0121
Record Dates: First submitted 2019-07-12; First posted 2019-07-15 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Eczema; MTOROC1 Signaling
Keywords: Eczema; MTORC1 Signaling; CBM Complex
MeSH Terms: conditions — Eczema | interventions — Glutamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): All patients will receive L-glutamine 10-30mg daily based on weight for 3 months
  Interventions: Drug: L-glutamine

INTERVENTIONS:
Drug: L-glutamine — product will be obtained by Endari and administered by NIH pharmacy. Patient will take supplement as prescribed

SUMMARY:
Background:

Glutamine is an amino acid. People get amino acids from food or from the body s cells. The body needs amino acids to stay healthy. Glutamine might help treat some people with immune system problems like atopic dermatitis.

Objective:

To study the safety and effectiveness of glutamine supplements for people with certain immune system problems.

Eligibility:

People ages 5-65 with atopic dermatitis and other immune system problems

Design:

Participants will be screened in another protocol.

Participants will have 8 visits.

Visit 1 includes:

Physical exam

Medical history

Blood and urine tests

Saliva sample

Nutrition assessment

For participants with AD, photographs of the skin

Participants will get a diary to record their symptoms every day during the study. They will record any glutamine side effects and bring the diary to every visit.

Visit 2 is about 1 month after visit 1. Participants will repeat visit 1 tests and get glutamine to take home. It is a powder that can be added to drinks or food. They will take it twice a day for 3 months. They will record their doses in a diary each day and bring the diary to all visits.

Participants will have a phone call 5 days after starting glutamine to discuss how they are feeling.

Visit 3 is about 7 days after participants start taking glutamine. They will have blood tests.

Visits 4, 5, and 6 occur each month participants are taking glutamine. Participants will repeat visit 1 tests.

Participants will stop taking glutamine after visit 6.

Visits 7 and 8 occur 1 and 3 months after participants stop taking glutamine. Participants will repeat visit 1 tests.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic, relapsing, inflammatory skin condition that typically begins in infancy or early childhood and can be highly debilitating with a marked reduction in quality of life. Current treatment modalities for AD include frequent use of skin moisturizers such as creams or emollients, topical corticosteroids and topical calcineurin inhibitors, systemic immunosuppressive drugs, and, in select cases of refractory disease, wet wrap therapy. The available systemic treatments for AD when topical treatment fails can have substantial adverse effects and are not always effective. The search for targeted therapies based on pathway disruptions in patients could present opportunities to provide therapies on a more personalized basis, tailored to the pathogenic pathways.

Based on prior studies, we have demonstrated that supplemental glutamine has potential as an effective AD treatment in patients with caspase activation and recruitment domain (CARD) gene mutations. Prior studies have demonstrated that loss of CARD signaling leads to a decrease in the mammalian target of rapamycin complex 1 (mTORC1) signaling pathway. Glutamine supplementation can normalize this defect in mTORC1. The CARD11 BCL10 MALT1 (CBM) signalosome complex is a critical component of mTORC1 activation. Some patients with gene mutations affecting the CBM complex do not develop AD but do develop other symptoms of immunoregulation and may also benefit from glutamine supplementation. We will conduct a phase 1, open-label study to investigate the use of supplemental glutamine in patients with immune dysregulation. Subjects 5 to 65 years of age will take oral glutamine daily for 3 months. To assess the role of the mTORC1 pathway in response to glutamine supplementation, we will enroll 3 groups of patients: 1) those with AD and a defect in mTORC1 signaling or a mutation in the CBM complex; 2) those with AD who do not have a defect in mTORC1 signaling or a mutation in the CBM complex; and 3) those who have a defect in mTORC1 signaling or a mutation in the CBM complex and do not have AD. Subjects will complete a daily symptom diary for 1 month before starting glutamine to document baseline disease status. Disease severity will be assessed at baseline, at the end of glutamine supplementation, and 1 and 3 months after completing the glutamine regimen. Blood will be collected periodically for safety, tolerability, and research assessments.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Be 5 to 65 years of age, inclusive.
* Able to provide informed consent.
* Be enrolled on NIAID protocol 10-I-0148 and identified on that protocol as meeting at least one of the following 3 criteria:

  * Has active, moderate-to-severe AD (defined as objective SCORAD greater than or equal to 15 or total SCORAD greater than or equal to 25).
  * Has a confirmed defect in mTORC1 signaling (based on T cell stimulation assay).
  * Has a confirmed CBM loss-of-function gene mutation (identified by genetic sequencing and verified in vitro by testing patient cells and/or transfection of mutant gene into cell lines).
* Females of childbearing potential must agree to use adequate contraception when engaging in sexual activities that can result in pregnancy, beginning 30 days prior to day 0 through study day 120. Acceptable methods of contraception include the following:

  * Continuous hormonal contraception used per label without interruption throughout the above period.
  * Male or female condom with spermicide.
  * Diaphragm or cervical cap with a spermicide.
  * Intrauterine device.
* Be willing to allow storage of biological samples for future research purposes.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Current, active infection requiring treatment.
* Current treatment with a chemotherapeutic agent.
* Participation in an ongoing research protocol evaluating an investigational agent.
* Treatment with approved prescription medications may be exclusionary, to be determined on a case-by-case basis by the principal investigator.
* Significant liver or kidney disease (serum glutamic oxaloacetic transaminase [SGOT], serum glutamine pyruvic transaminase [SGPT], or alkaline phosphatase >2.5 (SqrRoot) upper limit of normal [ULN], total bilirubin >1.5 (SqrRoot) ULN, or serum creatinine >1.5 (SqrRoot) ULN) in the past 30 days.
* Persons with an active seizure disorder. For persons with a prior history of seizures, the person should be seizure free for 5 years and not on any anti-seizure medication in order to be enrolled into the study. (Since glutamine is metabolized to glutamate and ammonia, and glutamate is the main excitatory neurotransmitter in the central nervous system, there is a theoretical increased risk of seizures.)

  * Allergy to monosodium glutamate.
  * Malabsorption.
  * Pregnancy.
  * Breastfeeding.
  * Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-12 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of glutamine supplementation in patients with immune disregulation. | 1 year
  assess safety and tolerability of glutamine

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Milner, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0121.html